CLINICAL TRIAL: NCT06460987
Title: Study of the Clinical Efficacy and Safety of Finerenone for the Treatment of IGA
Brief Title: Study of the Clinical Efficacy and Safety of Finerenone for the Treatment of IGA Nephropathy
Status: Completed | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2024-081
Record Dates: First submitted 2024-05-28; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Finerenone; IgA Nephropathy; Proteinuria; Safety Issues
Keywords: finerenone; IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — finerenone; Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A group: FINE+RASI group;: Patients treated with RASI and finerenone
  Interventions: Drug: Finerenone; Drug: RAS inhibitor
- B group: RASI group;: Patients treated with RASI only
  Interventions: Drug: RAS inhibitor
- C group: immune suppressive + FINE + RASI;: Patients receiving immunosuppressive drugs and RASIs
  Interventions: Drug: Finerenone; Drug: RAS inhibitor; Drug: Immune Suppressant
- D group: immune suppressive + RASI;: Patients receiving immunosuppressants, RASI and finerenone
  Interventions: Drug: RAS inhibitor; Drug: Immune Suppressant

INTERVENTIONS:
Drug: Finerenone — Taking the maximum tolerated dose of finerenone based on serum creatinine and blood potassium levels
  Other Names: FINE
  Groups: A group: FINE+RASI group;; C group: immune suppressive + FINE + RASI;
Drug: RAS inhibitor — Receive RAS inhibitor treatment as specified in the KDIGO guidelines
  Other Names: RASI
Drug: Immune Suppressant — Receive immune suppressant treatment as specified in the KDIGO guidelines
  Other Names: immunosupressive
  Groups: C group: immune suppressive + FINE + RASI;; D group: immune suppressive + RASI;

SUMMARY:
IgA nephropathy accounts for about 45 per cent of primary glomerular diseases in China and about 26 per cent of renal biopsies in patients with chronic failure.According to current guideline recommendations, there are limited indications for non-steroidal MRAs. Therefore clinical studies to explore the range of clinical indications for fenetyllone are warranted.

DETAILED DESCRIPTION:
Primary IgA nephropathy (IgAN) is an immunopathological diagnostic term for a type of glomerulonephritis characterised by the deposition of IgA or IgA-dominant immune complexes in the glomerular tunica albuginea. And in China IgA nephropathy accounts for about 45% of primary glomerular diseases and about 26% of renal biopsies in patients with chronic failure. Among them, about 15-40% of IgA nephropathy patients progress to renal failure after 10-20 years; IgA nephropathy has become one of the main causes of end-stage renal failure.The nonsteroidal salicorticoid receptor antagonist (MRA)- finerenone reduces the risk of composite renal outcomes, ESKD, or renal death in patients with type 2 diabetes and CKD.There are limited indications for non-steroidal MRAs. Therefore clinical studies to explore the range of clinical indications for fenetyllone are warranted.

ELIGIBILITY:
Inclusion Criteria:

* primary IgAN diagnosed by renal biopsy;
* receive RASI inhibitors for at least 3 months;
* serum potassium <5 mmol/L;
* protein-to-creatinine ratio (PCR) >0.3 mg/g

Exclusion Criteria:

* secondary IgAN;
* autosomal dominant polycystic kidney disease or autosomal recessive polycystic kidney disease, lupus nephritis, lupus nephritis,;
* previous renal transplantation;
* chronic hepatic disease, malignant tumor, active malignancy, heart failure with ejection fraction <40%;
* followed up less than 6 months;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IGA nephropathy by renal biopsy who met the inclusion exclusion criteria, were able to be followed up regularly, and had clinical follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
percentage change in PCR from baseline to 6 months | 6 month
  Collect PCR data before enrolment and at month 6 and calculate the percentage change

SECONDARY OUTCOMES:
percentage change in PCR from baseline to 1, 2 and 3 months | 1, 2 and 3 month
  Collec PCR before enrolment and at months 1, 2 and 3, then calculate the percentage change
frequency of patients with a 30% and 50% decrease in PCR | 6 month
  Calculate the number of patients with >30% or >50% reduction in proteinuria during the 6-month follow-up period
the level of change in eGFR | 6 month
  Collection of eGFR before enrolment and at months 6
the level of change in blood sodium | 6 month
  Collection of blood sodium before enrolment and at months 6
the level of change in serum creatinine | 6 month
  Collection of serum creatinine before enrolment and at months 6
the level of change in albumin | 6 month
  Collection of albumin before enrolment and at months 6

CONTACTS AND LOCATIONS:
Overall Officials: Qiaorui Wang, bachelor, Principal Investigator — Student
Locations (1):
- Study of the Clinical Efficacy and Safety of Finerenone for the Treatment of IGA Nephropathy, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang QR, Wu L, Huang J, Pan H, Wang XF, Li L, Han F, Wang YF, Wu ML, Yang Y. Efficacy and safety of finerenone in IgA nephropathy: an observational multicentre study. Clin Kidney J. 2025 Apr 28;18(5):sfaf125. doi: 10.1093/ckj/sfaf125. eCollection 2025 May. PMID 40357496

DOCUMENTS (1):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT06460987/Prot_000.pdf